CLINICAL TRIAL: NCT03852641
Title: Feeding Very-low-birth-weight (VLBW) Premature Infants (<1500g) During Non-invasive Respiratory Support- Continuous Drip Vs. Bolus Gavage Feeding
Brief Title: Feeding Premature Infants During Non-invasive Respiratory Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Liron Borenstein MD, Principal investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Feeding on NIPPV
Record Dates: First submitted 2019-02-20; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Premature Infant; Non-invasive Respiratory Support
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus gavage feeds (Experimental): Bolus gavage feeds over 15-30 minutes
  Interventions: Other: Length of feeding
- Continuous feeds (Experimental): Continuous feeds over 2.0 hrs
  Interventions: Other: Length of feeding

INTERVENTIONS:
Other: Length of feeding — Feeds will be given via nasogastric tube over 15-30 min versus 2 hr

SUMMARY:
A randomized control trial comparing bolus gavage feeds to continuous feed among premature infants supported by non-invasive respiratory support

ELIGIBILITY:
Inclusion Criteria:

* Infants <1500gr, on non-invasive respiratory support
* Feeding>20 ml/kg/day

Exclusion Criteria:

* Major congenital malformations
* Unstable infants because of sepsis, central nervous system, cardiac or other significant morbidities
* Gastrointestinal morbidity such as spontaneous intestinal perforation (SIP) and necrotising enterocolitis (NEC).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Oxygenation instability as documented by oxygen saturation histograms | before dischatge home at an average of 40 weeks gestation
Time to full feeds (TFF) defined as full enteral gavage feeding of 150 cc/Kg/day | before dischatge home at an average of 40 weeks gestation

SECONDARY OUTCOMES:
Respiratory-length of respiratory support | before dischatge home at an average of 40 weeks gestation
Incidence of Necrotising enterocolitis (NEC) as defined by the medical team | before dischatge home at an average of 40 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Liron Borenstein-Levin, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No